CLINICAL TRIAL: NCT06650670
Title: Randomized, Double-blind, Controlled Nutritional Intervention Study of Parallel Groups to Evaluate the Effect of Consuming a Bioactive Compound (EPP) on Joint Health in Healthy Adults
Brief Title: Effect of Consuming a Bioactive Compound (EPP) on Joint Health in Healthy Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of the strategic interest because the market potential is insufficient
Sponsor: Biosearch S.A. (Industry)
Collaborators: Universidad de Granada (Other); University Hospital Virgen de las Nieves (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C030
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Knee Discomfort
Keywords: extract; bioactive compound
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Control group that will receive two capsules with the maltodextrin per day during 12 weeks
  Interventions: Dietary Supplement: Dietary Supplement: Placebo
- EPP group (Experimental): Experimental group that will receive two capsules with the bioactive compound per day during 12 weeks
  Interventions: Dietary Supplement: Dietary Supplement: EPP

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Placebo — Each participant will consume 2 capsules per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: Control group
Dietary Supplement: Dietary Supplement: EPP — Each participant will consume 2 capsules per day in one of the main meals without any restriction in the diet or in their life habits
  Arms: EPP group

SUMMARY:
The objective of this trial is to determine the efficacy of oral administration of a bioactive compound (EPP) in healthy individuals with mild knee joint discomfort.

DETAILED DESCRIPTION:
It is estimated that the incidence of osteoarthritis (OA) is increasing exponentially worldwide, with serious consequences, not only on the quality of life and functionality of the subjects, but also a high burden on the social and health care systems of the countries. Existing treatments for OA are either invasive, and therefore risky for the subject and high cost, or have side effects and cannot be maintained over time. Therefore, there is a high demand to find effective and safe therapies to prevent and/or treat OA, such as functional ingredients or compounds present in food. In this regard, our experimental bioactive compound has been developed and shown to be safe and effective in reducing joint pain and improving quality of life in a previous study.

The aim of this study is to evaluate the effect of the consumption of our bioactive compound, in healthy Spanish individuals with mild joint discomfort in the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants (men and women) between 35 and 65 years of age with knee discomfort.
2. Mild knee joint pain (visual analog scale between 3 and 6 cm).

Exclusion Criteria:

1. People with clinical osteoarthritis or any other degenerative joint disease.
2. Persons receiving treatment with anti-inflammatory or chondroprotective drugs (chondroitin sulfate, glucosamine, HA, diacerein) two weeks prior to screening.
3. Persons receiving intra-articular injections in the knee joint in the 3 months prior to the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
KOOS test total score. | 12 weeks
  Using of the KOOS (Knee Injury & Osteoarthritis Outcomes) Questionnaire.

SECONDARY OUTCOMES:
KOOS Subscales score (pain, symptoms, daily activity, sport and quality of life). | 12 weeks
  Using the KOOS (Knee Injury & Osteoarthritis Outcomes) Questionnaire.
VPS scale for knee pain (general and after physical tests performed at the visits). | 12 weeks
  Using a Visual Pain Scale for Knee Pain
Objective assessment of physical activity. | 12 weeks
  The mobility of your knee will be assessed with a goniometer, the sit-to-stand test will be performed, and accelerometers will be collected to assess physical activity and sedentary lifestyle.
Range of motion of the knee joint. | 12 weeks
  The mobility of your knee will be assessed with a goniometer, the sit-to-stand test will be performed, and accelerometers will be collected to assess physical activity and sedentary lifestyle.
Changes observed between baseline and final MRI. | 12 weeks
  Analyzing cartilage by MRI
Lower body strength and power. | 12 weeks
  The mobility of your knee will be assessed with a goniometer, the sit-to-stand test will be performed, and accelerometers will be collected to assess physical activity and sedentary lifestyle.

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Ruiz Ruiz, Dr., Principal Investigator — Universidad de Granada
Locations (1):
- Universidad de Granada (Dpto. educación Física y Deportiva), Granada, Spain